CLINICAL TRIAL: NCT06576037
Title: Phase Ib Study of CBP-1019 in Combination With FOLFOX +/- Bevacizumab, Pembrolizumab, or Enzalutamide for Metastatic TRPV6-overexpressing Solid Tumors of Epithelial Origin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0474; NCI-2024-07312 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab; pembrolizumab; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part 1A: Dose Escalation CBP-1019 + FOLFOX (Experimental): Participants will be administered the study treatments on an outpatient basis.
  Interventions: Drug: CBP-1019; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-FLUOROURACIL
- Part 1B: Dose Escalation CBP-1019 + FOLFOX + Bevacizumab (Experimental): Participants will be administered the study treatments on an outpatient basis.
  Interventions: Drug: CBP-1019; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-FLUOROURACIL; Drug: Bevacizumab
- Part 1C: Dose Escalation CBP-1019 + Pembrolizumab (Experimental): Participants will be administered the study treatments on an outpatient basis.
  Interventions: Drug: CBP-1019; Drug: Pembrolizumab
- Part 1D: Dose Escalation CBP-1019 + Enzalutamide (Experimental): Participants will be administered the study treatments on an outpatient basis.
  Interventions: Drug: CBP-1019; Drug: Enzalutamide
- Part 2A: Pancreatic CBP-1019 + FOLFOX (Experimental): Participants will be administered the study treatments on an outpatient basis.
  Interventions: Drug: CBP-1019; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-FLUOROURACIL
- Part 2B: Colorectal CBP-1019 + FOLFOX + Bevacizumab (Experimental): Participants will be administered the study treatments on an outpatient basis.
  Interventions: Drug: CBP-1019; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-FLUOROURACIL; Drug: Bevacizumab
- Part 2C: Epithelial Origin CBP-1019 + Pembrolizumab (Experimental): Participants will be administered the study treatments on an outpatient basis.
  Interventions: Drug: CBP-1019; Drug: Pembrolizumab
- Part 2D: CRPC CBP-1019 + Enzalutamide (Experimental): Participants will be administered the study treatments on an outpatient basis.
  Interventions: Drug: CBP-1019; Drug: Enzalutamide

INTERVENTIONS:
Drug: CBP-1019 — Given by vein (IV)
Drug: Oxaliplatin — Given by vein (IV)
  Arms: Part 1A: Dose Escalation CBP-1019 + FOLFOX; Part 1B: Dose Escalation CBP-1019 + FOLFOX + Bevacizumab; Part 2A: Pancreatic CBP-1019 + FOLFOX; Part 2B: Colorectal CBP-1019 + FOLFOX + Bevacizumab
Drug: Leucovorin — Given by vein (IV)
  Arms: Part 1A: Dose Escalation CBP-1019 + FOLFOX; Part 1B: Dose Escalation CBP-1019 + FOLFOX + Bevacizumab; Part 2A: Pancreatic CBP-1019 + FOLFOX; Part 2B: Colorectal CBP-1019 + FOLFOX + Bevacizumab
Drug: 5-FLUOROURACIL — Given by vein (IV)
  Arms: Part 1A: Dose Escalation CBP-1019 + FOLFOX; Part 1B: Dose Escalation CBP-1019 + FOLFOX + Bevacizumab; Part 2A: Pancreatic CBP-1019 + FOLFOX; Part 2B: Colorectal CBP-1019 + FOLFOX + Bevacizumab
Drug: Bevacizumab — Given by vein (IV)
  Arms: Part 1B: Dose Escalation CBP-1019 + FOLFOX + Bevacizumab; Part 2B: Colorectal CBP-1019 + FOLFOX + Bevacizumab
Drug: Pembrolizumab — Given by vein (IV)
  Arms: Part 1C: Dose Escalation CBP-1019 + Pembrolizumab; Part 2C: Epithelial Origin CBP-1019 + Pembrolizumab
Drug: Enzalutamide — Given by mouth
  Arms: Part 1D: Dose Escalation CBP-1019 + Enzalutamide; Part 2D: CRPC CBP-1019 + Enzalutamide

SUMMARY:
An open-label, Phase Ib dose escalation and dose expansion clinical trial evaluating the safety and efficacy of CBP-1019 combinations in patients with solid tumors of epithelial origin.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the safety and tolerability of CBP-1019 combinations (Regimen A: CBP-1019 plus FOLFOX; Regimen B: CBP-1019 plus FOLFOX with bevacizumab; Regimen C: CBP-1019 plus pembrolizumab; and Regimen D: CBP-1019 plus enzalutamide) in metastatic solid tumors of epithelial origin.

To determine the ORR of CBP-1019 combinations in selected metastatic solid tumors of epithelial origin.

Secondary Objective:

To evaluate other indicators of the antitumor activity of CBP-1019 combinations.

Exploratory Objectives:

To explore potential biomarkers associated with response/resistance and major clinical outcomes (toxicity and antitumor activities) through molecular profiling at the DNA, RNA and protein levels.

To explore patient-reported outcomes (PROs).

ELIGIBILITY:
Inclusion Criteria

1. Patients must have histologically or cytologically confirmed malignancy of epithelial origin other than ovarian cancer that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective. Patients must have received at least one prior line of systemic standard therapy, and have either disease progression or intolerable toxicity after standard treatment.
2. In the dose expansion, Regimen A will enroll patients with metastatic pancreatic cancer with concurrent oxaliplatin and irinotecan-free interval ≥4 months (Cohort 1), Regimen B will enroll patients with metastatic colorectal cancer concurrent oxaliplatin and irinotecan-free interval ≥4 months (Cohort 2), Regimen C will enroll patients with metastatic solid tumors of epithelial origin who have received prior anti-PD-(L)1 therapy (Cohort 3), and Regimen D will enroll patients with metastatic castration-resistant and taxane-treated prostate cancer (Cohort 4).
3. Patients (with the exception of those with prostate cancer) must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥10 mm (≥1 cm) with computed tomography (CT) scan,PET-CT, magnetic resonance imaging (MRI) scan, or calipers by clinical exam.

   Note: Prostate cancer patients must meet ≥1 of the following Prostate Cancer Clinical Trials Working Group 3 criteria [95]:
   * Progression in measurable disease.
   * Bone disease progression defined by the appearance of ≥2 new bone lesions.
   * Prostate-specific antigen (PSA) progression defined as ≥2 sequential rises in PSA obtained ≥1 week apart with a minimal starting value of ≥1 ng/mL. A PSA value ≥2 ng/mL is required at study entry.
4. Ability to understand and the willingness to sign a written informed consent document.
5. Age ≥18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1 (Appendix 1).
7. Must have adequate organ and marrow functions as defined below:

   * Absolute neutrophil count (ANC) ≥1.5× 109/L: growth factor support is not allowed within 2 weeks of study treatment initiation.
   * Hemoglobin ≥9 g/dL: packed RBC transfusion is allowed as long as there is no active bleeding.
   * Platelets ≥100× 109/L: transfusion is not allowed within 2 weeks of study treatment initiation.
   * Total bilirubin ≤1.5× upper limit of normal (ULN); or total bilirubin <3.0× ULN with direct bilirubin ≤ ULN in patients with well documented Gilbert's syndrome.
   * Alanine aminotransferase (ALT) and AST ≤2.5× the upper limit of the reference range, or ≤ 5× the upper limit of the reference range for patients with liver metastases.
   * Serum albumin ≥3 g/dL.
   * Urinalysis ≤1 proteinuria, or urine protein/creatinine ratio (UPCR) ≤1 mg/mg (≤113.2 mg/mmol), or 24-h urine protein ≤1 g (applies to bevacizumab-based regimen only).
   * Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) ≤1.5× ULN if not on therapeutic anticoagulation.
   * Calculated creatinine clearance (CrCl) ≥50 mL/min by the Cockcroft-Gault method as below or 24-hour urine collection.

CrCl = (140-age) × (weight/kg) x Fa / (72 × serum creatinine mg/dL). a where F= 0.85 for females and F=1 for males 9. Patients whose baseline pulse oximetry is at least 90% on room air.

10. Fridericia's corrected QT interval (QTcF =QT/∛(60/HR) ) ≤460 ms for males and ≤480 ms for females on electrocardiogram (ECG) conducted at rest during screening.

Note: Patients with an atrioventricular pacemaker or other condition (e.g., right bundle branch block) that renders the QT measurement invalid are an exception and this criterion does not apply.

11. The effects of study drugs on the developing human fetus are unknown. For this reason and because Class II drugs as well as other therapeutic agents used in this trial are known to be teratogenic, women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, throughout the study treatment period, and for 6 months after study treatment completion (Refer to Pregnancy Assessment Policy MDACC Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (follicle-stimulating hormone and estradiol in menopausal range and have received whole pelvic radiation therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device (IUD), tubal ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

  12. Females of childbearing potential must have a negative serum pregnancy test within 3 days prior to study treatment initiation (Cycle 1 Day 1).

  13. Men and women enrolled on this protocol must agree to use adequate contraception during the study treatment period and for 6 months after completion of study treatment.

  14. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimens are eligible for this trial.
* Agree to provide baseline tumor specimens: archival tissue block, or 10 FFPE slides, or a pre-treatment biopsy.
* Patients must have adequate washout from prior therapy at the time of study treatment initiation: 3 weeks from any treatment specifically for systemic tumor control; 2 weeks from cytotoxic agents that were administered weekly; 6 weeks from nitrosoureas or mitomycin C; and 5 half-lives from targeted agents with half-lives and pharmacodynamic effects lasting <5 days.

Exclusion Criteria

1. Has received an investigational non-myelosuppressive agent within 14 days prior to study treatment initiation or an investigational myelosuppressive agent within 21 days prior to study treatment initiation.
2. Uncontrolled intercurrent illness including but not limited to:

   * Ongoing or active infection requiring IV antibiotics.
   * Symptomatic congestive heart failure (New York Heart Association Class III or IV).
   * History of myocardial infarction, unstable angina, stroke, or transient ischemic attack within 6 months before study enrollment.
   * Lesions invading or encasing any major blood vessels and cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation; uncontrolled hypertension defined as sustained blood pressure >140 mmHg systolic / >90 mmHg diastolic despite optimal antihypertensive treatment (applies to bevacizumab-based regimen only).
   * History or current evidence of uncontrolled ventricular arrhythmia.
   * Congenital long QT syndrome, or any known history of torsade de pointes, or family history of unexplained sudden death.
   * Clinically significant bleeding or active gastric or duodenal ulcer.
   * Chronic diarrhea disease considered to be clinically significant by the investigator.
   * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before the first dose of study treatment, or any GI disorders associated with a high risk of perforation or fistula formation.
   * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

   Note: Patients with a diagnosis of incidental subsegmental pulmonary embolism or deep vein thrombosis are allowed if stable, asymptomatic, and on a stable dose of anticoagulant for at least 1 week before the first dose of study treatment.
3. Unresolved clinically significant Grade ≥1 toxicity from prior therapy. Note: Patients who were exposed to prior treatment with any of the combination regimens that experienced intolerable or severe toxicity, even if they recovered; or who required dose reduction of chemotherapy or enzalutamide in their standard of care therapies should be excluded.
4. History of allergic reactions to the study drugs or any of their components.
5. Has not recovered from a major surgical procedure or significant traumatic injury (i.e., still needing additional surgical or medical care for these issues): major surgical procedures ≤28 days prior to study entry or minor surgical procedures ≤7 days prior to study entry. No waiting period is required following port-a-cath or other central venous access placement. Patients must have complete wound healing from major or minor surgery before the first dose of study treatment.
6. Currently receiving an investigational drug in a clinical trial or participating in any other type of medical research judged not to be scientifically or medically compatible with this study. If a patient is currently enrolled in a clinical trial involving non-approved use of a therapeutic device for cancer control, then agreement with the investigator and the Sponsor is required to establish eligibility.
7. Has received a live vaccine within 30 days prior to the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: Bacille Calmette-Guérin vaccine, measles, mumps, rabies, rubella, typhoid vaccine, varicella/zoster, and yellow fever. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed. COVID-19 vaccines including killed virus are allowed.
8. Symptomatic primary tumors or metastasis in the brain and/or central nervous system (CNS) that are uncontrolled with antiepileptics and/or require prednisone >10 mg/day or equivalent.

   Note: Patients with treated brain metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no evidence of progression. Patients with asymptomatic, new, or progressive brain metastases (active brain metastases) are eligible if the treating physician determines that immediate CNS-specific treatment is not required and is unlikely to be required during the first cycle of study treatment.
9. Evidence of leptomeningeal or lymphangitic carcinomatosis.
10. Patients with a history of stem cell or solid organ transplantation.
11. Breastfeeding or pregnant.
12. Known history of positive test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).

    Patients with a history of positive HIV test result who meet all the following eligibility criteria may be enrolled:
    * Have a T cell (CD4+) count ≥350 cells/μL.
    * No history of opportunistic infections or other malignancies.
    * Have an HIV viral load less than 400 copies/mL.
    * In the opinion of the investigator, their antiretroviral therapy or other HIV treatments will not interfere with the activity of the investigational product or cause any confusion with the assessment of the investigational drug toxicities.

    Patients with a history of positive HBV or HCV test result must have:
    * Negative viral load test (HBV DNA or HCV RNA) at screening.
13. Ability to take oral medications without medical history of malabsorption or other chronic GI disease, or other conditions that may hamper compliance and/or absorption of the study agent (applies to enzalutamide-based regimen only).
14. Concurrent immunosuppressive therapy or steroid therapy (>10 mg/day prednisone or equivalent) (applies to pembrolizumab-based regimen only).
15. History of autoimmune disease including but not limited to inflammatory bowel disease, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis that required systemic therapy in the past 2 years (applies to pembrolizumab-based regimen only).

    Note: Patients with vitiligo, resolved childhood asthma/atopy, hypothyroidism on stable hormone replacement, controlled asthma, type I diabetes, Graves' disease, or Hashimoto's disease are not excluded.
16. History of Grade ≥2 immune related reactions (i.e., uveitis, etc.) that prompted prior immune checkpoint inhibitor therapy discontinuation (applies to pembrolizumab-based regimen only).

    Note: Patients with adequately treated skin rash other than Steven-Johnson syndrome, toxic epidermal necrolysis, or other severe forms of dermatitis and patients on replacement therapy for endocrinopathies are not excluded (applies to pembrolizumab-based regimen only).
17. History of interstitial lung disease or (non-infectious) pneumonitis that required steroids or current pneumonitis (applies to pembrolizumab-based regimen only).
18. History of Grade ≥3 allergic reaction to treatment with a monoclonal antibody (applies to bevacizumab-based and pembrolizumab-based regimens only).
19. Patients who experienced oxaliplatin-related Grade 3 peripheral neuropathy or any grade neuropathy that triggered oxaliplatin discontinuation (applies to FOLFOX-based regimens only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org